CLINICAL TRIAL: NCT01795638
Title: Impact of Early Postnatal Sodium Supplementation on Weight Gain in Very Low Birth Weight Infants
Brief Title: Sodium Supplementation and Growth in Very Low Birth Weight Infants
Acronym: SSALT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The unit's standard nutrition practices change which impacted our methodology.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 09-07-28-07
Record Dates: First submitted 2013-02-13; First posted 2013-02-21 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2016-03

CONDITIONS: Extreme Immaturity
Keywords: anthropometrics; weight; nutrition
MeSH Terms: conditions — Body Weight | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium chloride (Active Comparator): Sodium chloride 1 meq/kg (0.4 ml/kg of 2.5meq/ml formulation for injection)q6hrs on days of life 7-35. Intervention was given enterally if feedings were at least 100 ml/kg/day; otherwise medication was diluted in equal amounts of dextrose 5% water and administered intravenously.
  Interventions: Drug: Sodium chloride
- sterile water (Placebo Comparator): Sterile water, 0.4 ml/kg q6hrs on days of life 7-35. Placebo is given enterally when infant is tolerating at least 100 ml/kg/day; otherwise the product is diluted in equal amounts of dextrose 5% water and administered intravenously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium chloride
  Arms: Sodium chloride
Drug: Placebo — sterile water, 0.4 ml/kg every 6 hours on days of life 7-35.
  Other Names: Sterile Water
  Arms: sterile water

SUMMARY:
Adequate growth during the neonatal period is critical for optimal long term outcomes. Despite maximal calorie intake, sixty percent of very low birth weight infants still fail to thrive suggesting that factors other than total calorie intake are important in ensuring consistent weight gain. Several reports have indicated a positive sodium balance is critical in ensuring good weight gain in very low birth weight infants, however these infants are susceptible to low serum sodium concentrations. Urine sodium values are sometimes used to diagnosis of hyponatremia or negative sodium balance after the first two weeks of life, but there is no evidence for this practice in preterm neonates. Our central hypothesis is that early supplementation with sodium will ensure positive sodium balance in very low birth weight infants and will result in optimal weight gain and enhanced long term outcomes. Secondarily we hypothesize that low sodium concentrations in the urine will not correlate with low serum sodium values.

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled trial in infants born at less than 32 weeks gestation, who are admitted to the Newborn Intensive Care Unit at University of Cincinnati Medical Center, Cincinnati, Ohio. Infants are randomized to receive either 4 meq/kg/day supplemental sodium or an equal amount of sterile water on days of life 7-35. Institutional data from 2008 revealed that a sample size of 56 infants completing the study will detect a 15% difference in the primary outcome of weight gain with 80% power and an alpha error of 0.05. Allowing that 33% drop-out rate (infants may be transferred to another hospital, expire, or be discharged prior to day of life 35), we choose to randomize 75 infants. Calorie intake, serum sodium, weight gain, urine sodium were monitored weekly till 35 days of life or discharge. Infants were assessed for common morbidities associated with prematurity including bronchopulmonary dysplasia, systemic hypertension, late-onset sepsis, necrotizing enterocolitis and retinopathy of prematurity.

ELIGIBILITY:
Inclusion Criteria:

* infants born at less than 32 weeks postmenstrual age

Exclusion Criteria:

* infants with major malformations deemed incompatible with life disease states characterized by edema renal failure, defined as an increase in serum creatinine by 0.5 mg/dl/day or urine output less than 0.5 ml/kg/hour

Ages: 7 Days to 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry T Akinbi, MD, Study Director — Cincinnati Childrens Hospital Medical Center
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Sodium chloride 1 meq/kg (0.4 ml/kg of 2.5meq/ml formulation for injection)q6hrs on days of life 7-35. Intervention was given enterally if feedings were at least 100 ml/kg/day; otherwise medication was diluted in equal amounts of dextrose 5% water and administered intravenously.
  Sodium chloride
- Placebo: Sterile water, 0.4 ml/kg q6hrs on days of life 7-35. Placebo is given enterally when infant is tolerating at least 100 ml/kg/day; otherwise the product is diluted in equal amounts of dextrose 5% water and administered intravenously.
  Placebo: sterile water, 0.4 ml/kg every 6 hours on days of life 7-35.
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 27 | 26
Completed | 14 | 15
Not Completed | 13 | 11
Not completed — Death | 0 | 3
Not completed — transferred to quaternary hospital | 2 | 3
Not completed — Protocol Violation | 3 | 0
Not completed — discharged from hospital | 7 | 5
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Infants met inclusion criteria and [parents consented for their infants to participate
Groups:
- Sodium Chloride: Sodium chloride 1 meq/kg (0.4 ml/kg of 2.5meq/ml formulation for injection)q6hrs on days of life 7-35. Intervention was given enterally if feedings were at least 100 ml/kg/day; otherwise medication was diluted in equal amounts of dextrose 5% water and administered intravenously.
  Sodium chloride
- Total: Total of all reporting groups
Arm/Group | Sodium Chloride | Sterile Water | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Median (Full Range); unit: weeks] | 28.4 [24 to 31.9] | 29.3 [23.9 to 31.7] | 28.5 [24 to 31.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 13 | 11 | 24
Weight at birth in grams [Median (Full Range); unit: grams] | 1080 [551 to 1669] | 1021 [551 to 1785] | 1051 [551 to 1785]
Body length at birth in centimeters [Median (Full Range); unit: centimeters] | 35.8 [27 to 41] | 34.9 [28.5 to 39] | 35.4 [27 to 41]
Head circumference at birth in centimeters [Median (Full Range); unit: centimeters] | 25.1 [21.5 to 29] | 24.6 [21.5 to 28] | 24.9 [21.5 to 29]
Modified CRIB score [Median (Full Range); unit: units on a scale] — Clinical Risk Index for Babies scoring system (CRIB II) score is a tool to predict initial risk of mortality amongst low birth weight babies.
  Scale ranges: 0-15 with 0 being the least severe and 15 being the most severe
  units on a scale | 1 [0 to 15] | 2 [0 to 15] | 1 [0 to 15]
Maternal Milk as Primary Diet [Number; unit: participants] | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain at Six Weeks of Age
Description: Average weight gain in g/kg/day and also as a % birthweight over the first six weeks of the study will be compared between the two study arms
Time Frame: Six weeks of age
Measure: Median (Inter-Quartile Range); unit: g/kg/day
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 14 | 15
g/kg/day | 26.9 [24.7 to 29.2] | 22.4 [20.2 to 24.6]

2. Secondary Outcome: Body Length at Six Weeks of Age
Description: The percentage of infants maintaining birth percentile at six weeks between the two study arms will be analyzed
Time Frame: six weeks of age
Measure: Number; unit: percentage
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 14 | 15
percentage | 14 | 15

3. Secondary Outcome: Head Circumference
Description: The percentage of infants maintaining birth percentile for head circumference will be compared between the two groups.
Time Frame: six weeks of age
Measure: Number; unit: percent
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 14 | 15
percent | 14 | 15

4. Secondary Outcome: Mean Systolic Blood Pressure
Description: Systolic blood pressures at 36 weeks post-conceptual age will be compared between the two groups
Time Frame: 36 weeks post-conceptual age
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 14 | 15
mmHg | 84.4 [74 to 96] | 81.8 [70 to 90]

5. Secondary Outcome: Chronic Diuretic Therapy
Description: The incidence of chronic diuretic therapy will be compared between the two groups
Time Frame: patients will be followed during birth hospital stay; an expected average of 3 months of age
Measure: Number; unit: participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 14 | 15
participants | 4 | 3

6. Secondary Outcome: Late-onset Sepsis
Description: The incidence of late-onset sepsis, defined as positive blood culture for credible pathogen and/or 5 days of continuous antimicrobial therapy after the first week of life will be compared between the two groups.
Time Frame: patients will be followed during birth hospitalization; an expected average of 3 months of age
Measure: Number; unit: participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 27 | 26
participants | 2 | 12

7. Secondary Outcome: Necrotizing Enterocolitis
Description: The incidence of Bell stage II or greater necrotizing enterocolitis after the second week of life will be compared between the two groups
Time Frame: patients will be followed during birth hospitalization; an expected average of 3 months of age
Measure: Number; unit: participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 27 | 26
participants | 0 | 4

8. Secondary Outcome: Chronic Lung Disease
Description: The incidence of chronic lung disease, defined as respiratory support at 36 weeks postmenstrual age will be compared between the two groups
Time Frame: 36 weeks post-mentrual age
Measure: Number; unit: participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 27 | 26
participants | 9 | 5

9. Secondary Outcome: Mortality
Description: The incidence of death during birth hospitalization will be compared between the two study arms
Time Frame: patients will be followed during birth hospitalization; an expected 3 months of age
Measure: Number; unit: participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 27 | 26
participants | 0 | 4

10. Secondary Outcome: Patent Ductus Arteriosus
Description: prolonged Patent Ductus Arteriosus after the second week of life
Time Frame: After the second week of life
Measure: Number; unit: participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 27 | 26
participants | 7 | 9

ADVERSE EVENTS:
Arm/Group | Intervention | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 3/27 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=27) | Placebo (N=26)
hypernatremia (Metabolism and nutrition disorders) | 3 | 0 — three infants receiving intervention contemporaneously with maintainence intravenous fluids developed hypernatremia (range 150-151mmol/L) and were withdrawn from the study, per defined protocol.

LIMITATIONS AND CAVEATS:
Study was terminated after 95% of sample size was recruited. Small number of subjects are analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No